CLINICAL TRIAL: NCT05144854
Title: A Randomized, Multicenter, Open-label, Phase III Study to Compare the Efficacy and Safety of ONO-4538 in Combination With Ipilimumab, Fluoropyrimidine-based and Platinum-based Chemotherapy (Hereinafter Referred to as "Chemotherapy") Versus Chemotherapy in Chemotherapy-naïve Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Negative Unresectable Advanced or Recurrent Gastric Cancer (Including Esophagogastric Junction Cancer)
Brief Title: A Study to Evaluate the Efficacy and Safety of ONO-4538 in Combination With Ipilimumab and Chemotherapy in Chemotherapy-naïve Participants With HER2-negative Unresectable Advanced or Recurrent Gastric Cancer (Including Esophagogastric Junction Cancer)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4538-113
Record Dates: First submitted 2021-10-06; First posted 2021-12-03 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Nivolumab; Ipilimumab; Oxaliplatin; Capecitabine; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ONO-4538 + ipilimumab + chemotherapy (Experimental)
  Interventions: Drug: ONO-4538; Drug: Ipilimumab; Drug: Oxaliplatin; Drug: Capecitabine; Drug: S-1
- Chemotherapy (Active Comparator)
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: S-1

INTERVENTIONS:
Drug: ONO-4538 — Specified dose on specified days
  Other Names: Nivolumab; Opdivo
  Arms: ONO-4538 + ipilimumab + chemotherapy
Drug: Ipilimumab — Specified dose on specified days
  Other Names: BMS-734016; Yervoy
  Arms: ONO-4538 + ipilimumab + chemotherapy
Drug: Oxaliplatin — Specified dose on specified days
Drug: Capecitabine — Specified dose on specified days
Drug: S-1 — Specified dose on specified days
  Other Names: Tegafur-gimeracil-oteracil potassium

SUMMARY:
This study is to compare and evaluate the efficacy and safety of ONO-4538 in combination with ipilimumab and chemotherapy versus chemotherapy in chemotherapy-naïve participants with HER2-negative unresectable advanced or recurrent gastric cancer (including esophagogastric junction cancer).

ELIGIBILITY:
Inclusion Criteria:

1. Participants with unresectable advanced or recurrent gastric cancer (including esophagogastric junction cancer) that has been histologically confirmed to be predominant adenocarcinoma
2. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score 0 or 1
3. Participants who have a life expectancy of at least 3 months

Exclusion Criteria:

1. Participants with a history or complications of multiple cancers
2. Participants with a complication or history of severe hypersensitivity to any other antibody products
3. Participants with concurrent autoimmune disease or a history of chronic or recurrent autoimmune disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | up to 3 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) (site investigator assessment) | up to 3 years
Objective response rate (ORR) (site investigator assessment) | up to 3 years
Best overall response (BOR) (site investigator assessment) | up to 3 years
Duration of response (DOR) (site investigator assessment) | up to 3 years
Disease control rate (DCR) (site investigator assessment) | up to 3 years
Time to response (TTR) (site investigator assessment) | up to 3 years
Maximum percent change in the sum diameters of the target lesions (site investigator assessment) | up to 3 years
Progression-free survival after the next line of therapy (PFS2) (site investigator assessment) | up to 3 years
Adverse event | Up to 30 days after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (57):
- Japan (12):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Osaki Citizen Hospital, Osaki-shi, Miyagi
  - Osaka University Hospital, Suita-shi, Osaka
  - Saitama Medical University International Medical Center, Hidaka-shi, Saitama
  - Saitama Cancer Center, Ina-machi, Kitaadati-gun, Saitama
  - Shizuoka Cancer Center, Nagaizumi-Cho, Sunto-Gun, Shizuoka
  - University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - IMSUT Hospital, The Institute of Medical Science, The University of Tokyo, Minato-ku, Tokyo
  - Keio University Hospital, Shinjyuku-ku, Tokyo
- South Korea (29):
  - Kosin University Gospel Hospital, Busan, Gangwon-do
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Kyungpook National University Chilgok Hospital, Daegu, Gyeongsangbuk-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Jeonbuk national university hospital, Jeonju, Jeollabuk-do
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Dong-A University Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Konyang University Hospital, Daejeon
  - Gachon University Gil Medical Center, Incheon
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Taiwan (16):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital, Keelung, Keelung
  - Far Eastern Memorial Hospital, New Taipei City
  - Taipei Medical University - Shuang Ho Hospital, Ministry of Health and Welfare, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Hospital, Liouying, Tainan
  - National Cheng Kung University Hospital, Tainan
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Municipal Wanfang Hospital Managed by Taipei Medical University, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital,Linkou, Taoyuan

IPD SHARING:
Plan to Share IPD: No